CLINICAL TRIAL: NCT00220558
Title: A Randomized Comparison of Sirolimus Eluting Stent Versus Bare Metal Stent in Chronic Total Coronary Occlusions: The Gruppo Italiano di Studio Sullo Stent Nelle Occlusioni Coronariche. The GISSOC II Study.
Brief Title: GISSOC II: Sirolimus Eluting Stent Versus Bare Metal Stent in Chronic Total Coronary Occlusions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Società Italiana di Cardiologia Invasiva (Other)
Collaborators: Cordis Italy a division of Johnson & Johnson Medical SpA (Unknown)
Responsible Party: Dr. Paolo Rubartelli, Ospedale Villascassi, Genova Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRDIT 00-01/04
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Transluminal Coronary Angioplasty; Bare metal stents; drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Coronary placement of bare metal stent vs. drug eluting stent

SUMMARY:
The objective of this study is to compare the Cypher Select-TM Sirolimus Eluting Stent (SES) with the SONIC-TM Bare Metal Stent (BMS) in the treatment of Chronic Total Occlusion lesions (CTO). The primary hypothesis is that, at 8-month follow-up, the minimal luminal diameter (MLD) of the coronary segment treated with stent implantation in CTO lesions is significantly larger with the use of SES compared to BMS. The treated segment is defined as the segment covered by the stent(s) plus 5 mm proximally and distally to the stent(s).

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized study that will be conducted at up to 22 centers in Italy. All patients who meet the eligibility criteria will be randomized to Cypher Select-TM Stent or SONIC-TM Stent. Patients will have repeat angiography at 8 months and clinical follow-up to 2 years. The study population will consist of 150 patients with single chronic total occlusion in a native coronary artery with a reference diameter between 2.75 mm and 3.75 mm. The occlusion has to be dilatable by balloon angioplasty and can be fully covered by < 2 stents of ≤33 mm of length each. The CTO is defined as obstruction of a native coronary artery, at least 30 days old, with no luminal continuity and with Thrombolysis in Myocardial Infarction (TIMI) flow grade 0 or 1. Following confirmation of eligibility criteria and successful pre-dilating of the CTO, patients will be randomized in a 1:1 ratio to receive SES CYPHER SELECT Stent or BMS SONIC Stent.

The coronary angiograms will be assessed at a core laboratory with Quantitative Coronary Angiography. Quantitative angiographic parameters including minimal luminal diameter, binary restenosis rate, total reocclusion rate, late luminal loss, will be evaluated at 8 months. The incidence of clinical events, including death, myocardial infarction, target vessel revascularization, stent thrombosis, will be evaluated at 8, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable angina pectoris or documented silent ischemia;
* Planned treatment of a single de novo chronic totally occluded (CTO) in a native coronary artery with a reference diameter between 2.75 mm and 3.75 mm;
* The target lesion can be fully covered by ≤ 2 stents of ≤33 mm of length each;
* The target CTO is at least 30 days old;
* The target CTO is successfully crossed by a guide wire and dilated by a balloon;

Exclusion Criteria:

* Myocardial infarction within 30 days in the territory of the target CTO;
* Unprotected left main coronary artery disease;
* Target CTO is in a graft;
* Target CTO is in a stented segment;
* Presence of other lesions in the same vessel,requiring angioplasty and not treatable with the same stent(s) used for the target CTO;
* More than one CTO requiring PCI;
* Target CTO has diseased side branches >2.0 mm in diameter;
* Target CTO pretreated with non-balloon devices such as atherectomy or laser or thrombectomy devices;
* Patient treated with coronary brachytherapy;
* The patient has an ejection fraction ≤ 30%;
* The patient has impaired renal function (creatinine > 3.0 mg/dl);
* The patient has known allergies to aspirin, clopidogrel bisulfate and ticlopidine, heparin, or sirolimus, contrast media or stainless steel that cannot be managed medically;
* The patient needs therapy with warfarin;
* The patient has a life expectancy less than 24 months;
* Recipient of heart transplant;
* The patient is currently participating in an investigational drug or another device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-05; Primary Completion 2007-10 (Actual); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
The minimal luminal diameter (MLD) at 8-month follow-up of the coronary segment treated with stent implantation in CTO lesions. The treated segment is defined as the segment covered by the stent(s) plus 5 mm proximally and distally to the stent(s). | 8 month

SECONDARY OUTCOMES:
- Major adverse cardiac events (MACE) rate at 30 days, 8, 12 and 24 months; | two years
- In-segment late loss (LL) at 8 months; | 8 months
- Binary restenosis rate in the treated coronary segment, defined as the rate of patients showing an in-segment diameter stenosis greater than 50% at 8 months; | eight month
- In-segment total re-occlusion at 8 months; | 8 month
- Target Lesion Revascularization (TLR) at 8 ,12 and 24 months; | two years
- Target Vessel Revascularization (TVR) at 8 ,12 and 24 months; | two years
- Angiographic success defined as achievement of a final residual diameter stenosis of < 30 % (by QCA)using the assigned study stent; | procedure date
- Procedural success defined as angiographic success, without the occurrence of death, myocardial infarction (MI), or repeat revascularization of the target lesion during the hospital stay; | procedure date
- Sub acute stent thrombosis defined as angiographic documentation <30 days after the index procedure (site-reported or by QCA) of thrombus or total occlusion at the target site and freedom from an interim revascularization of the target vessel; | one month
- Late stent thrombosis defined as angiographic documentation >30 days after the index procedure (site-reported or by QCA) of thrombus or total occlusion at the target site and freedom from an interim revascularization of the target vessel. | two yeras

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rubartelli, MD, Principal Investigator — Azienda Ospedaliera Villa Scassi - Genoa - Italy
Locations (14):
- Italy (14):
  - Ospedale San Donato, Arezzo
  - Cliniche Gavazzeni, Bergamo
  - Ospedale Sant'Orsola-Malpighi, Bologna
  - Ospedale Vittorio Emanuele, Catania
  - Ospedale Sant'Anna, Como
  - Azienda Ospedaliera Villa Scassi, Genoa
  - Ospedale San Martino, Genova
  - Ospedale Civile di Legnano, Legnano
  - Ospedale Civile di Mestre, Mestre
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Pisana, Pisa
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale San Giovanni Battista Università, Torino
  - Ospedale Cà Foncello, Treviso

REFERENCES:
- [Background] Rubartelli P, Niccoli L, Verna E, Giachero C, Zimarino M, Fontanelli A, Vassanelli C, Campolo L, Martuscelli E, Tommasini G. Stent implantation versus balloon angioplasty in chronic coronary occlusions: results from the GISSOC trial. Gruppo Italiano di Studio sullo Stent nelle Occlusioni Coronariche. J Am Coll Cardiol. 1998 Jul;32(1):90-6. doi: 10.1016/s0735-1097(98)00193-4. PMID 9669254
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Hoye A, Tanabe K, Lemos PA, Aoki J, Saia F, Arampatzis C, Degertekin M, Hofma SH, Sianos G, McFadden E, van der Giessen WJ, Smits PC, de Feyter PJ, van Domburg RT, Serruys PW. Significant reduction in restenosis after the use of sirolimus-eluting stents in the treatment of chronic total occlusions. J Am Coll Cardiol. 2004 Jun 2;43(11):1954-8. doi: 10.1016/j.jacc.2004.01.045. PMID 15172397
- [Derived] Rubartelli P, Petronio AS, Guiducci V, Sganzerla P, Bolognese L, Galli M, Sheiban I, Chirillo F, Ramondo A, Bellotti S; Gruppo Italiano di Studio sullo Stent nelle Occlusioni Coronariche II GISE Investigators. Comparison of sirolimus-eluting and bare metal stent for treatment of patients with total coronary occlusions: results of the GISSOC II-GISE multicentre randomized trial. Eur Heart J. 2010 Aug;31(16):2014-20. doi: 10.1093/eurheartj/ehq199. Epub 2010 Jun 20. PMID 20566487
- See also: Società Italiana di Cardiologia Invasiva — http://www.gise.it/